CLINICAL TRIAL: NCT03076320
Title: Molecular and Clinical Study of the Effect of Zaxcell Versus Effezel in the Inflammatory and Scarring Process of Moderate and Severe Acne
Brief Title: Pirfenidone Plus M-DDO Gel in Moderate and Severe Acne
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Civil de Guadalajara (Other); Cell Pharma (Other)
Responsible Party: Principal Investigator, Juan Armendáriz-Borunda, PhD, FAASLD, Director of Institute of Molecular Biology in Medicine, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBMMTG 15-02; 008/16 (Other: Hospital Civil de Guadalajara Investigative Committee); 267/15 (Other: Hospital Civil de Guadalajara Etical of Investigative Committee)
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Acne Vulgaris Superficial Mixed Comedonal and Inflammatory
Keywords: Modified diallyl disulfide oxide (M-DDO); Pirfenidone (PFD); Adapalene + Benzoyl peroxide (A-BPO)
MeSH Terms: interventions — Pyridones; Adapalene; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFD+M-DDO (Experimental): Pirfenidone with M-DDO Active ingredients: Pirfenidone 10% with modified oxide diallyl disulfide (M-DDO) 0.016% Dosage form: gel. Dosage: standard finger tip unit (0.5g for an area of 100 to 120 square centimeters).
  Frequency an duration: topically applied every 12 hours for 6 months.
  Interventions: Combination Product: PDF+M-DDO
- A+PBO (Active Comparator): Adapalene with benzoyl peroxide Active ingredients: 0.1% Adapalene with 2.5% benzoyl peroxide. Dosage form: gel. Dosage: standard finger tip unit (0.5g for an area of 100 to 120 square centimeters).
  Frequency and duration: topically applied every 12 hours for 6 month
  Interventions: Combination Product: A+PBO

INTERVENTIONS:
Combination Product: PDF+M-DDO — Participants with moderate and severe acne will be treated two times a day on the face and superior back with a smooth layer (standard finger tip unit 0.5 g for an area of 100 to 120 square centimeters) of Zaxcell (Pirfenidone with M-DDO) in form of a gel. Patients have to wait 20 min without cover those sites.
  Other Names: Zaxcell; 5-methyl-phenyl-2(1h)- pyridone with M-DDO
  Arms: PFD+M-DDO
Combination Product: A+PBO — Participants with moderate and severe acne will be treated once a day (at night) on the face and superior back with a smooth layer (standard finger tip unit 0.5 g for an area of 100 to 120 square centimeters) of Effezel (Adapalene with benzoyl peroxide) in form of a gel. Patients have to wait 20 min without cover those sites
  Other Names: Effezel; Adapalene with benzoyl peroxide
  Arms: A+PBO

SUMMARY:
Acne vulgaris is a complex skin disorder involving multiple abnormalities of the pilosebaceous unit. Acne is the most common skin disease during puberty and worsens throughout adolescence. However, epidemiological studies suggest that acne can arise at any age, most frequently affecting individuals between puberty and 30 years of age, with 79%-95% of subjects aged between 16 years and 18 years and 80% of subjects between puberty and 30 years of age. Acne is considered the main reason for consultation with the dermatologist in institutional and private clinical practice.

Clinical features include seborrhoea, non-inflammatory lesions, inflammatory lesions and various degrees of scarring. There are many classifications of acne and scarring severity. Moderate to severe acne is about 15-20%.

Facial acne scarring affects both sexes equally and occurs to some degree in up to 95% of cases. There is a significant correlation between the initial acne grade and the overall severity of scarring at all sites and in both sexes. This would suggest that treatment aimed at reducing the severity of acne might reduce the incidence of scarring. Both superficial inflammatory acne lesions as well as deep nodular lesions seem capable of producing scars.

Conventional therapies recommended for the treatment of acne vulgaris include retinoids, benzoyl peroxide (BPO), antibiotics, and hormonal therapy. Combination therapy using agents with complementary mechanisms provides the opportunity to target multiple pathogenetic causes of acne vulgaris.

The combination in gel with 0.1% adapalene and 2.5% BPO is a once-daily treatment of acne vulgaris. In several double- blind, randomized controlled trials (RCTs), the Adapalene-BPO (A-BPO) combination therapy applied once daily for 12 weeks significantly reduced the number of both inflammatory and non-inflammatory lesions in subjects with moderate acne vulgaris. In Mexico there is an available commercial product of this combination (Effezel®; Galderma). The limitation of this topical therapy is the low tolerability by patients as they can experiment several levels of irritation, erythema, dryness, desquamation, burning, and itching), and patients are advised to expect these side effects, which contribute to discontinue therapy if it becomes severe.

On the other hand, 5-methyl-1-phenyl-2-(1h)-pyridone or pirfenidone (PFD) is a wide-spectrum antifibrotic drug that modulates diverse cytokines action, involving TGF-β, TNF-α, epidermal growth factor, platelet-derived growth factor, VEGF, IGF-1, fibroblast growth factor, interferon-γ, interleukin (IL)-1, IL-6, and IL-8 and it has shown promising effects in vitro and in vivo settings. Also, PFD has proven effective in the prevention and regression of pulmonary fibrosis, peritoneal sclerosis, hepatic cirrhosis, uterine fibromyoma, left ventricular fibrosis, renal interstitial fibrosis, and breast capsular contracture in experimental models. A recently open phase II clinical trial evaluated the therapeutic use of PFD gel in localized scleroderma. Results showed it acts on both the inflammatory and the fibrotic phases.

The other component of Zaxcell is modified-diallyl disulfide oxide (M-DDO) an antimicrobial and antiseptic agent, which has been proved in patients with chronic diabetic ulcer as a potent germicide and has show to increase the beneficial effect of PFD preventing infections, accelerating and improving ulcer resolution. (Observations not published).

According to this, the investigators believe that Zaxcell (PFD + M-DDO) could play an important role in the modulation of inflammatory and scarring process in acne. The investigators hypothesis is that PFD in patients with moderate to severe acne modulates amplification of the inflammatory response, regulating the inflammasome activation, macrophage polarization and its activity in regulating the wound healing process of the skin in an early fashion.

Zaxcell is an innovative gel with a synergetic mode of action that could modulate the inflammatory response. Furthermore, has antiseptic properties and regulates the process of wound healing, fibrogenic and scarring process. In vitro and in vivo studies provide an initial body of evidence on the safety and clinical benefits of PFD, the main component of Zaxcell as a promising candidate for the treatment of moderate to severe acne.

DETAILED DESCRIPTION:
Participants will be randomized using a random number table to distribute in the control (Effezel) and the experimental group (Pirfenidone+M-DDO). Before screening, participants will undergo an informed consent process and they will sign an institutional review board-approved informed consent form. The study will be conducted in accordance with Good Clinical Practices and the principles that have their origins in the Declaration of Helsinki (revised Seoul, Korea, 2008). Potential subjects with acne scars will be selected from the investigators practices and solicited from advertisements. To be included, subjects must have met the inclusion criteria. Demographics data and medical history will be registered on a monthly basis. Before treatment, all subjects with inflammation and scars will be evaluated in the face and back area using the Investigator´s Global Assessment scale (IGA scale) and all the lesions will be counted. The face and back area affected will be mapped and photographed. Participants in the experimental group will receive topical Zaxcell (Pirfenidone 10% +M-DDO gel) two times a day on the face and superior back and patients in control group will receive Effezel (Adapalene 0.1%+Benzoyl peroxide 2.5%) once a day. Both groups will apply the topical treatment in acne on the face and superior back area for six months previous cleansing of the area with neutral soap. Two biopsies of skin will be taken at the beginning, at month one and month 3 from the back area where the treatment will be applied. After this time, only clinical evaluations and photographs will be performed. Participants will be evaluated at every month until 6 months after their last application.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders male or female of any race, 12 to 25 years or age.
* Subjects with a clinical diagnosis of acne vulgaris with facial and back involvement.
* Subjects with a minimum of 20 but not more tan 150 inflammatory lesions on the face (including the nose)
* Subjects with a minimum of 30 but no more 200 non-inflammatory lesions on the face (including the nose)
* Subjects with minimum of 20 but no more than 250 inflammatory lesions on the superior back area.
* Investigator's Global Assessment (IGA) score of 3 or 4, corresponding to moderate and severe acne. Subjects with no more than two active nodules at baseline.
* Subjects that agree to fill a clinical history, access to physical exploration and biochemical analysis samples, biopsy of the back and photo-documentation of affected areas on the face and back.
* Consent to participate, verified by signing an approved written Informed Consent Form, or for subjects under age 18, an assent form in conjunction with a signed Informed Consent Form from a parent/guardian.
* Patients willing to sign a compliance letter to apply treatment as indicated by the principal investigator.
* Willingness and capacity of protocol compliance (for subjects under 18 years of age, parent/guardian must be wiling and able to comply with study requirements).
* Subjects willing to share personal information and data as verified by signing a written authorization, as applicable

Exclusion Criteria:

* Acne conglobata, acne fulminans, secondary acne.
* Subjects with another chronic inflammatory disease of the skin.
* Subjects with severe acne requiring isotretinoin therapy or other dermatological conditions, which might, in the opinion of the Investigator, interfere with the study evaluation or pose a risk to patient safety during the study.
* Pregnancy, nursing or planning a pregnancy.
* Men with facial hair that would interfere with the assessments.
* Subjects with background history of keloid scarring.
* Known sensitivities to the study preparations.
* Participation in another investigational drug or device research study within 30 day of enrollment.
* Specified washout period to baselines for systemic or topical medications.
* Subjects refusing to the biopsy of the back and photographic procedures.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Assessing change of lesions with IGA scale (Investigators' Global Assessment) | 1, 2, 3, 4, 5 and 6 months
  Number or lesions

SECONDARY OUTCOMES:
Histopathological modification on the inflammatory lesions and improvement in the scarring process | 1 and 3 months
  Biopsy from the upper back area
2. Expression levels of key molecules involved in acne inflammation and scar remodeling | 1 and 3 months
  Biopsy from the upper back area
Photonumeric scale | 1, 3 and 6 months
  Photographs of the treated area analyzed by three-dimensional reconstruction software

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Gollnick HP, Finlay AY, Shear N; Global Alliance to Improve Outcomes in Acne. Can we define acne as a chronic disease? If so, how and when? Am J Clin Dermatol. 2008;9(5):279-84. doi: 10.2165/00128071-200809050-00001. PMID 18717602
- [Background] Kang S, Cho S, Chung JH, Hammerberg C, Fisher GJ, Voorhees JJ. Inflammation and extracellular matrix degradation mediated by activated transcription factors nuclear factor-kappaB and activator protein-1 in inflammatory acne lesions in vivo. Am J Pathol. 2005 Jun;166(6):1691-9. doi: 10.1016/s0002-9440(10)62479-0. PMID 15920154
- [Background] Macias-Barragan J, Sandoval-Rodriguez A, Navarro-Partida J, Armendariz-Borunda J. The multifaceted role of pirfenidone and its novel targets. Fibrogenesis Tissue Repair. 2010 Sep 1;3:16. doi: 10.1186/1755-1536-3-16. PMID 20809935
- [Background] Zhou R, Jiang X. Effects of adapalene-benzoyl peroxide combination gel in treatment or maintenance therapy of moderate or severe acne vulgaris: a meta-analysis. Ann Dermatol. 2014 Feb;26(1):43-52. doi: 10.5021/ad.2014.26.1.43. Epub 2014 Feb 17. PMID 24648685
- [Background] Rodriguez-Castellanos M, Tlacuilo-Parra A, Sanchez-Enriquez S, Velez-Gomez E, Guevara-Gutierrez E. Pirfenidone gel in patients with localized scleroderma: a phase II study. Arthritis Res Ther. 2015 Jan 28;16(6):510. doi: 10.1186/s13075-014-0510-4. PMID 25533576
- [Background] Holland DB, Jeremy AH. The role of inflammation in the pathogenesis of acne and acne scarring. Semin Cutan Med Surg. 2005 Jun;24(2):79-83. doi: 10.1016/j.sder.2005.03.004. PMID 16092795